CLINICAL TRIAL: NCT04417569
Title: A Proof of Concept Study to Determine the Rise of Progesterone Levels After Human Chorionic Gonadotrophin (hCG) Trigger in Stimulated Cycles of IVF/ICSI
Brief Title: A Proof of Concept Study of Serum Progesterone Levels for IVF/ICSI Following HCG Trigger for Oocyte Maturation
Status: Completed | Type: Observational
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Sponsor
Other Study IDs: 2002-ABU-001-CC
Record Dates: First submitted 2020-05-18; First posted 2020-06-04 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Infertility; Infertility, Female; IVF; hCG
MeSH Terms: conditions — Infertility; Infertility, Female | interventions — Chorionic Gonadotropin; Ultrasonography; Hematologic Tests; Progesterone; Luteinizing Hormone; Estradiol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- stimulated cycles: Patients will have blood drawn on five separate occasions: before and following hCG trigger on the day of final oocyte maturation and day of egg collection
  Interventions: Drug: hCG; Diagnostic Test: Ultrasound; Other: Blood test

INTERVENTIONS:
Drug: hCG — human chorionic gonadotropin
  Other Names: human chorionic gonadotropin
Diagnostic Test: Ultrasound — Endometrial thickness monitoring
  Other Names: transvaginal scan
Other: Blood test — Progesterone, Luteinizing Hormone, Estradiol
  Other Names: Progesterone, Luteinizing Hormone, Estradiol

SUMMARY:
This study will determine the rise of progesterone levels after human chorionic gonadotrophin (hCG) trigger in stimulated cycles IVF/ICSI

DETAILED DESCRIPTION:
Studies have suggested that controlled ovarian hyperstimulation adversely affects endometrial receptivity. In ovarian stimulation cycles with exogenous gonadotrophins there is an ongoing debate regarding the effect of a late follicular phase progesterone level on reproductive outcomes. It is not yet clarified if an elevated serum progesterone level in the late follicular phase is a symptom or cause of an adverse effect on reproductive outcomes. A new hypothesis is evolving and gaining momentum providing a novel explanation for the association between late follicular phase progesterone rise and reproductive outcome. It is proposed that exogenous FSH (Follicle-stimulating hormone) administration results in supraphysiological levels of FSH, which induce an abundance of LH (luteinizing hormone) receptors on granulosa cells causing the follicles to become hypersensitive to LH-like activity (ie hCG trigger). Based on this hypothesis, the focus should be placed on the hCG trigger rather than on the late follicular phase progesterone rise.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18 to 42 years with regular menstrual cycles of 26-34 days
* Undergoing ovarian stimulation for IVF/ICSI & PGS.
* Receiving recombinant FSH for stimulation
* hCG 5000iu IM as trigger injection for oocyte maturation.
* Ovarian stimulation in GnRH-antagonist protocols
* BMI 18- 35 kg/m2
* Having 1 or 2 euploid embryos for transfer in spontaneous natural cycles.

Exclusion Criteria:

* Poor ovarian reserve as defined by Bologna criteria
* PCOS in accordance with Rotterdam criteria

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Female patients who are planned to commence ovarian stimulation for IVF/ICSI with hCG trigger for oocyte maturation and plan to avail of pre-implantation genetic screening with embryo vitrification of their biopsied embryos at blastocyst stage
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Level of progesterone day of trigger | 1 day
  day of the hCG trigger between 1000h - 1200h, before trigger, 1 hour after trigger, 2 hrs after trigger

SECONDARY OUTCOMES:
Level of progesterone day of egg retrieval | 1 day
  36hrs after trigger

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Loja Vitorino, Specialist, Principal Investigator — ART Fertility Clinics LLC
Locations (1):
- ART Fertility Clinics LLC, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bourgain C, Devroey P. The endometrium in stimulated cycles for IVF. Hum Reprod Update. 2003 Nov-Dec;9(6):515-22. doi: 10.1093/humupd/dmg045. PMID 14714588
- [Result] Devroey P, Bourgain C, Macklon NS, Fauser BC. Reproductive biology and IVF: ovarian stimulation and endometrial receptivity. Trends Endocrinol Metab. 2004 Mar;15(2):84-90. doi: 10.1016/j.tem.2004.01.009. PMID 15036255
- [Result] Kolibianakis E, Bourgain C, Albano C, Osmanagaoglu K, Smitz J, Van Steirteghem A, Devroey P. Effect of ovarian stimulation with recombinant follicle-stimulating hormone, gonadotropin releasing hormone antagonists, and human chorionic gonadotropin on endometrial maturation on the day of oocyte pick-up. Fertil Steril. 2002 Nov;78(5):1025-9. doi: 10.1016/s0015-0282(02)03323-x. PMID 12413988
- [Result] Nikas G, Develioglu OH, Toner JP, Jones HW Jr. Endometrial pinopodes indicate a shift in the window of receptivity in IVF cycles. Hum Reprod. 1999 Mar;14(3):787-92. doi: 10.1093/humrep/14.3.787. PMID 10221715
- [Result] Simon C, Garcia Velasco JJ, Valbuena D, Peinado JA, Moreno C, Remohi J, Pellicer A. Increasing uterine receptivity by decreasing estradiol levels during the preimplantation period in high responders with the use of a follicle-stimulating hormone step-down regimen. Fertil Steril. 1998 Aug;70(2):234-9. doi: 10.1016/s0015-0282(98)00140-x. PMID 9696213
- [Result] Weinerman R, Mainigi M. Why we should transfer frozen instead of fresh embryos: the translational rationale. Fertil Steril. 2014 Jul;102(1):10-8. doi: 10.1016/j.fertnstert.2014.05.019. Epub 2014 Jun 2. PMID 24890274
- [Result] Liu Y, Lee KF, Ng EH, Yeung WS, Ho PC. Gene expression profiling of human peri-implantation endometria between natural and stimulated cycles. Fertil Steril. 2008 Dec;90(6):2152-64. doi: 10.1016/j.fertnstert.2007.10.020. Epub 2008 Jan 14. PMID 18191855
- [Result] Haouzi D, Assou S, Mahmoud K, Tondeur S, Reme T, Hedon B, De Vos J, Hamamah S. Gene expression profile of human endometrial receptivity: comparison between natural and stimulated cycles for the same patients. Hum Reprod. 2009 Jun;24(6):1436-45. doi: 10.1093/humrep/dep039. Epub 2009 Feb 26. PMID 19246470
- [Result] Roque M, Lattes K, Serra S, Sola I, Geber S, Carreras R, Checa MA. Fresh embryo transfer versus frozen embryo transfer in in vitro fertilization cycles: a systematic review and meta-analysis. Fertil Steril. 2013 Jan;99(1):156-162. doi: 10.1016/j.fertnstert.2012.09.003. Epub 2012 Oct 3. PMID 23040524
- [Result] Roque M, Valle M, Guimaraes F, Sampaio M, Geber S. Freeze-all policy: fresh vs. frozen-thawed embryo transfer. Fertil Steril. 2015 May;103(5):1190-3. doi: 10.1016/j.fertnstert.2015.01.045. Epub 2015 Mar 4. PMID 25747130
- [Result] Haas J, Smith R, Zilberberg E, Nayot D, Meriano J, Barzilay E, Casper RF. Endometrial compaction (decreased thickness) in response to progesterone results in optimal pregnancy outcome in frozen-thawed embryo transfers. Fertil Steril. 2019 Sep;112(3):503-509.e1. doi: 10.1016/j.fertnstert.2019.05.001. Epub 2019 Jun 24. PMID 31248618
- [Result] Testart J, Frydman R, Feinstein MC, Thebault A, Roger M, Scholler R. Interpretation of plasma luteinizing hormone assay for the collection of mature oocytes from women: definition of a luteinizing hormone surge-initiating rise. Fertil Steril. 1981 Jul;36(1):50-4. doi: 10.1016/s0015-0282(16)45617-7. PMID 7250407
- [Result] Irani M, Robles A, Gunnala V, Reichman D, Rosenwaks Z. Optimal parameters for determining the LH surge in natural cycle frozen-thawed embryo transfers. J Ovarian Res. 2017 Oct 16;10(1):70. doi: 10.1186/s13048-017-0367-7. PMID 29037231
- [Result] Groenewoud ER, Macklon NS, Cohlen BJ; ANTARCTICA Study Group. The effect of elevated progesterone levels before HCG triggering in modified natural cycle frozen-thawed embryo transfer cycles. Reprod Biomed Online. 2017 May;34(5):546-554. doi: 10.1016/j.rbmo.2017.02.008. Epub 2017 Feb 28. PMID 28319018
- [Result] Fatemi HM, Kyrou D, Bourgain C, Van den Abbeel E, Griesinger G, Devroey P. Cryopreserved-thawed human embryo transfer: spontaneous natural cycle is superior to human chorionic gonadotropin-induced natural cycle. Fertil Steril. 2010 Nov;94(6):2054-8. doi: 10.1016/j.fertnstert.2009.11.036. Epub 2010 Jan 25. PMID 20097333
- [Result] Bosch E, Labarta E, Crespo J, Simon C, Remohi J, Jenkins J, Pellicer A. Circulating progesterone levels and ongoing pregnancy rates in controlled ovarian stimulation cycles for in vitro fertilization: analysis of over 4000 cycles. Hum Reprod. 2010 Aug;25(8):2092-100. doi: 10.1093/humrep/deq125. Epub 2010 Jun 10. PMID 20539042
- [Result] Griesinger G, Mannaerts B, Andersen CY, Witjes H, Kolibianakis EM, Gordon K. Progesterone elevation does not compromise pregnancy rates in high responders: a pooled analysis of in vitro fertilization patients treated with recombinant follicle-stimulating hormone/gonadotropin-releasing hormone antagonist in six trials. Fertil Steril. 2013 Dec;100(6):1622-8.e1-3. doi: 10.1016/j.fertnstert.2013.08.045. Epub 2013 Sep 29. PMID 24083873
- [Result] Venetis CA, Kolibianakis EM, Bosdou JK, Tarlatzis BC. Progesterone elevation and probability of pregnancy after IVF: a systematic review and meta-analysis of over 60 000 cycles. Hum Reprod Update. 2013 Sep-Oct;19(5):433-57. doi: 10.1093/humupd/dmt014. Epub 2013 Jul 4. PMID 23827986
- [Result] Yding Andersen C, Bungum L, Nyboe Andersen A, Humaidan P. Preovulatory progesterone concentration associates significantly to follicle number and LH concentration but not to pregnancy rate. Reprod Biomed Online. 2011 Aug;23(2):187-95. doi: 10.1016/j.rbmo.2011.04.003. Epub 2011 Apr 28. PMID 21665546
- [Result] Friis Wang N, Skouby SO, Humaidan P, Andersen CY. Response to ovulation trigger is correlated to late follicular phase progesterone levels: A hypothesis explaining reduced reproductive outcomes caused by increased late follicular progesterone rise. Hum Reprod. 2019 May 1;34(5):942-948. doi: 10.1093/humrep/dez023. PMID 30927415
- [Derived] Coughlan C, Vitorino R, Melado L, Digma S, Sibal J, Patel R, Lawrenz B, Fatemi H. Evolution of serum progesterone levels in the very early luteal phase of stimulated IVF/ICSI cycles post hCG trigger: a proof of concept study. J Assist Reprod Genet. 2022 May;39(5):1095-1104. doi: 10.1007/s10815-022-02474-4. Epub 2022 Apr 7. PMID 35391631